CLINICAL TRIAL: NCT00469729
Title: A Multi-Center, Multi-National, Historical Cohort Controlled Study to Evaluate Efficacy and Safety of Transplantation of StemEx®, Umbilical Cord Blood Stem and Progenitor Cells Expanded Ex Vivo, in Subjects With Hematologic Malignancies Following Myeloablative Therapy
Brief Title: Efficacy and Safety Study of StemEx®, to Treat Subjects With High Risk Hematologic Malignancies, Following Myeloablative Therapy
Acronym: ExCell
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gamida Cell -Teva Joint Venture Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#02.01.001; NCT00763334 (obsolete NCT alias)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2013-03

CONDITIONS: Hematologic Malignancies; Acute Myeloid Leukemia; Lymphoid Leukemia; Chronic Myeloid Leukemia; Hodgkin's Disease; Non-Hodgkin's Lymphoma; Myelodysplastic Syndromes
Keywords: Tetraethylenepentamine; Umbilical Cord Blood Stem Cell Transplantation; Hematological Malignancies; Acute Lymphoid Leukemia; Subjects with high-risk hematologic malignancies who are candidates for allogeneic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Leukemia, Lymphoid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- StemEx (Experimental)
  Interventions: Drug: StemEx®

INTERVENTIONS:
Drug: StemEx® — The stem/progenitor cell based product composed of ex vivo expanded allogeneic umbilical cord blood cells, which is infused to subject at a rate of 1-3 ml/min in combination with non-manipulated cells derived from the same cord blood unit.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of transplanting StemEx® in patients with certain hematological malignancies. For these patients, it is suggested that StemEx® can improve upon the outcome of transplanting a single, unmanipulated cord blood unit by significantly increasing the number of stem/progenitor cells available to the patient.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation is a life-saving procedure for patients with hematologic malignancies; yet wide application of this procedure is limited by the availability of suitably Human Leukocyte Antigen (HLA) - matched donors. Only 30% of patients who could benefit from this procedure have an HLA-matched sibling. The lengthy search for a matched donor may critically delay transplantation. In addition, far fewer patients of racial minorities find suitable HLA-matched donors. Umbilical cord blood (UCB) has been increasingly used as an alternative source of stem cells; however, its use in adults and adolescent patients is limited due to insufficient cell dose required for satisfactory hematopoietic reconstitution.

Gamida Cell - Teva Joint Venture Ltd. is engaged in the development of StemEx®, an expanded hematopoietic UCB stem cell graft, as a potential medicinal product for the treatment of cancer and hematological malignancies. The expansion technology enables preferential expansion of hematopoietic stem and early progenitor cells and is based on the findings that copper chelators can regulate the balance between self-renewal and differentiation of stem cells.

The multi-national, multi-center Phase II/III clinical study designated to evaluate the safety and efficacy of StemEx® will enroll approximately 100 subjects with high-risk hematologic malignancies who are candidates for allogeneic stem cell transplantation (SCT). This study will evaluate the effect of StemEx® on overall survival as measured by overall 100-day mortality.

The study consists of 4 phases:

1. Screening phase includes subjects' clinical assessment and screening tests
2. Conditioning phase includes the myeloablative treatment prior transplantation procedure
3. Transplantation and post-transplant follow-up phase to day 180
4. Observational phase: survival status follow-up to day 730 (18 months)

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of AML or ALL: CR2 or subsequent complete remission (CR) or CR1 with high-risk features or relapse with < 10% blasts in BM and no circulating blasts.
2. Clinical diagnosis of CML: in CP1 (Chronic Phase 1) and resistant or intolerant to Gleevec or in CP2 or subsequent CP or in accelerated phase.
3. Clinical diagnosis of HD: induction failure or relapse and sensitive to last chemotherapy course.
4. Clinical diagnosis of NHL induction failure or relapse and sensitive to last chemotherapy course.
5. Clinical diagnosis of MDS with intermediate 2- or high-risk IPSS score.

Exclusion Criteria:

1. Less than twenty-one days have elapsed since the subject's last radiation or chemotherapy prior to conditioning (except Hydroxyurea).
2. HIV positive.
3. Pregnancy or lactation.
4. Uncontrolled bacterial, fungal or viral infection.
5. Subjects with signs and symptoms of active central nervous system (CNS) disease.
6. Availability of appropriate related and willing stem cell donor, who is HLA-matched at 5 or 6/6 antigens.
7. Prior allogeneic cell transplant.
8. Allergy to bovine or to any product, which may interfere with the treatment.
9. Enrolled in another clinical trial or received an investigational treatment during the last 30 days, unless approved by Sponsor.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2007-10; Primary Completion 2013-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall 100-day mortality | 100 days

SECONDARY OUTCOMES:
180 day mortality, acute Graft versus Host Disease (GvHD) grades III-IV, engraftment failure | 180 days
Safety and tolerability measures: The incidence and frequency of adverse experiences, acute toxicity, laboratory data and vital signs follow-up. | 180 days
Proportion of overall mortality at 1 year | One year post transplant
Proportion of overall mortality at 2 years | Two years post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wah Chan, MD, Principal Investigator — Texas Transplant Institute; Scott D Rowley, MD, Principal Investigator — The Cancer Center at Hackensack University Medical Center; Mary Territo, MD, Principal Investigator — UCLA Oncology Center; Patrick Stiff, MD, Principal Investigator — Loyola University Cardinal Bernardin Cancer Center; Agha Mounzer, MD, Principal Investigator — University of Pittsburgh Cancer Institute/UPMC Cancer Centers; Entezam Sahovic, MD, Principal Investigator — The Western Pennsylvania Hospital; Celia Grosskreutz, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Roger Giller, MD, Principal Investigator — The Children's Hospital, B115, University of Colorado Health Sciences Center; Steven Neudorf, MD, Principal Investigator — Children's Hospital of Orange County; Ronit Yerushalmi, MD, Principal Investigator — Chaim Sheba Medical Center; Tsila Zuckerman, MD, Principal Investigator — Rambam Health Care Campus; Christelle Ferra, MD, Principal Investigator — Germans Trias i Pujol Hospital; Cristina Arbona, MD, Principal Investigator — Hospital Clínico Universitario de Valencia; Guillermo Sanz, MD, Principal Investigator — Hospital Universitario La Fe; William Arcese, MD, Principal Investigator — Universita di Roma Tor Vergata; Alberto Bosi, MD, Principal Investigator — Ospedale di Careggi BMT Unit Department of Haematology; Sonali Chaudhury, MD, Principal Investigator — Northwestern University School of Medicine, Stem Cell Transplant Program, Children's Memorial Hospital; Jorge Sierra, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Igor B. Resnick, MD, PhD, Principal Investigator — Department of Bone Marrow Transplantation And Cancer Immunotherapy Hebrew University Hospital Ein-Karem, Jerusalem; Prof. Franco Locatelli, MD, Principal Investigator — Ospedale Pedriatrico Bambino Gesù; Dr. Mi Kwon, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón; Dr. Pere Barba, MD, Principal Investigator — Hospital Universitario Vall d´Hebrón; Dr. Cristina Diaz de Heredia, MD, Principal Investigator — Hospital Universitario Vall d´Hebrón; Prof. Mary J Laughlin, MD, Principal Investigator — Hematopoietic Stem Cell Transplant Program, University of Virginia
Locations (30):
- United States (16):
  - UCLA's Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - The Children's Hospital, B115, University of Colorado Health Sciences Center, Aurora, Colorado
  - Northwestern University School of Medicine, Stem Cell Transplant Program, Children's Memorial Hospital, Chicago, Illinois
  - Cardinal Bernardin Cancer Center, Loyola University Stritch School of Medicine, Maywood, Illinois
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cornell University, Joan & Sanford I. Weill Medical College, New York, New York
  - Steven and Alexandra Cohen Children's Medical Center of New York, New York, New York
  - Mount Sinai Medical Center, One Gustave L Levy Place, BOX 1410, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute/UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Texas Transplant Institute, San Antonio, Texas
  - University of Virginia, Hematopoietic Stem Cell Transplant Program, West Complex 1300 Jefferson Park Av, Charlottesville, Virginia
  - Medical College of Wisconsin Division of Neoplastic Diseases and Related Disorders, Milwaukee, Wisconsin
  - Medical College of Wisconsin Pediatric Blood and Marrow Transplant Program, Milwaukee, Wisconsin
- Szent Laszlo & Szent Istvan Hospital, Budapest, Hungary
- Israel (3):
  - Hebrew University Hospital Ein-Karem, Department of Bone Marrow Transplantation And Cancer Immunotherapy, Jerusalem
  - Rambam Medical Center, PO Box 9602, Haifa
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Ospedale Pedriatrico Bambino Gesù, Roma
  - Universita di Roma Tor Vergata, Via Oxford 81, Roma
  - Ospedale di Careggi BMT Unit Department of Haematology, Viale Morgagni, Florence
- Spain (7):
  - Hospital Clínico Universitario de Valencia, Avda. Blasco Ibañez, 17, Valencia, Valencia
  - Hospital Universitario La Fe, Av Campanar 21, Valencia
  - Hospital de la Santa Creu i Sant Pau, C/ Sant Antoni Maria Claret, Barselona
  - Hospital Germans Trias i Pujol, Carretera de Canyet S/n, Badalona
  - Hospital General Universitario Gregorio Marañón, Doctor Esquerdo 46 , Madrid
  - Hospital Universitario Vall d´Hebrón (Pediatrics), Passeig de La Vall d´Hebrón 119-129, Barcelona
  - Hospital Universitario Vall d´Hebrón, Passeig de La Vall d´Hebrón 119-129, Barcelona

REFERENCES:
- [Background] Peled T, Landau E, Prus E, Treves AJ, Nagler A, Fibach E. Cellular copper content modulates differentiation and self-renewal in cultures of cord blood-derived CD34+ cells. Br J Haematol. 2002 Mar;116(3):655-61. doi: 10.1046/j.0007-1048.2001.03316.x. PMID 11849228
- [Background] Peled T, Landau E, Mandel J, Glukhman E, Goudsmid NR, Nagler A, Fibach E. Linear polyamine copper chelator tetraethylenepentamine augments long-term ex vivo expansion of cord blood-derived CD34+ cells and increases their engraftment potential in NOD/SCID mice. Exp Hematol. 2004 Jun;32(6):547-55. doi: 10.1016/j.exphem.2004.03.002. PMID 15183895
- [Background] Prus E, Peled T, Fibach E. The effect of tetraethylenepentamine, a synthetic copper chelating polyamine, on expression of CD34 and CD38 antigens on normal and leukemic hematopoietic cells. Leuk Lymphoma. 2004 Mar;45(3):583-9. doi: 10.1080/10428190310001598035. PMID 15160922
- [Background] Peled T, Mandel J, Goudsmid RN, Landor C, Hasson N, Harati D, Austin M, Hasson A, Fibach E, Shpall EJ, Nagler A. Pre-clinical development of cord blood-derived progenitor cell graft expanded ex vivo with cytokines and the polyamine copper chelator tetraethylenepentamine. Cytotherapy. 2004;6(4):344-55. doi: 10.1080/14653240410004916. PMID 16146887
- [Background] Peled T, Glukhman E, Hasson N, Adi S, Assor H, Yudin D, Landor C, Mandel J, Landau E, Prus E, Nagler A, Fibach E. Chelatable cellular copper modulates differentiation and self-renewal of cord blood-derived hematopoietic progenitor cells. Exp Hematol. 2005 Oct;33(10):1092-100. doi: 10.1016/j.exphem.2005.06.015. PMID 16219531
- [Background] Shpall EJ, M.d.L., K. Chan, R. Champlin, A. Gee, P. Thall, K. Komanduri, D. Couriel, C. Hosing, B. Andersson, R. Jones, S. Giralt, S. Karandish, T. Sadeghi, B. Muriera, S. O'Connor, L. Wooten, X. Wang, S. Robinson, P. Fu, J. Wilson, T. Peled, F. Grynspan, A. Nagler, J. McMannis; A Phase I/II Study of Ex Vivo Expanded Cord Blood for Leukemia and Lymphoma. ISCT 2005 - conference publication, 2005.
- [Background] de Lima M, McMannis J, Gee A, Komanduri K, Couriel D, Andersson BS, Hosing C, Khouri I, Jones R, Champlin R, Karandish S, Sadeghi T, Peled T, Grynspan F, Daniely Y, Nagler A, Shpall EJ. Transplantation of ex vivo expanded cord blood cells using the copper chelator tetraethylenepentamine: a phase I/II clinical trial. Bone Marrow Transplant. 2008 May;41(9):771-8. doi: 10.1038/sj.bmt.1705979. Epub 2008 Jan 21. PMID 18209724
- [Derived] Stiff PJ, Montesinos P, Peled T, Landau E, Goudsmid NR, Mandel J, Hasson N, Olesinski E, Glukhman E, Snyder DA, Cohen EG, Kidron OS, Bracha D, Harati D, Ben-Abu K, Freind E, Freedman LS, Cohen YC, Olmer L, Barishev R, Rocha V, Gluckman E, Horowitz MM, Eapen M, Nagler A, Sanz G. Cohort-Controlled Comparison of Umbilical Cord Blood Transplantation Using Carlecortemcel-L, a Single Progenitor-Enriched Cord Blood, to Double Cord Blood Unit Transplantation. Biol Blood Marrow Transplant. 2018 Jul;24(7):1463-1470. doi: 10.1016/j.bbmt.2018.02.012. Epub 2018 Mar 1. PMID 29477778
- See also: Sponsor's website — http://www.gamida-cell.com/
- See also: Patients Against Lymphoma — http://www.lymphomation.org
- See also: Bone and Marrow Transplant Information Network — http://www.bmtinfonet.org/
- See also: NCI Leukemia Homepage — http://www.cancer.gov/cancertopics/types/leukemia
- See also: Leukemia information on MediciNet.com — http://www.medicinenet.com/leukemia/article.htm
- See also: American Society for Blood and Marrow Transplantation — http://www.asbmt.org/
- See also: American Society of Hematology — http://www.hematology.org/
- See also: Lymphoma Research Foundation — http://www.lymphoma.org
- See also: American Cancer Society website — http://www.cancer.org/docroot/home/index.asp
- See also: Center for International Blood and Marrow Transplant Research — http://www.cibmtr.org/
- See also: National Marrow Donor Program — http://www.marrow.org/
- See also: Children's Hospital of Orange County — http://www.choc.org/
- See also: University of Colorado Cancer Center — http://www.ucdenver.edu/academics/colleges/medicalschool/centers/cancercenter/Pages/CancerCenter.aspx
- See also: Northwestern University School of Medicine, Stem Cell Transplant Program, Children's Memorial Hospital website — http://www.childrensmemorial.org/depts/stemcell/overview.aspx
- See also: Duke University Medical Center — http://medschool.duke.edu/
- See also: Case Western Reserve University — http://www.case.edu/
- See also: University of Pittsburgh Cancer Institute — http://www.upmccancercenters.com/
- See also: MD Anderson Cancer Center — http://www.mdanderson.org/
- See also: Texas Transplant Institute — http://www.texastransplant.org/
- See also: Hôpital Saint Louis — http://www.chu-stlouis.fr/
- See also: Chaim Sheba Medical Center — http://eng.sheba.co.il/
- See also: Rambam Medical Center — http://www.rambam.org.il/
- See also: Universita di Roma Tor Vergata — http://web.uniroma2.it/home.php?sr=1024
- See also: Ospedale di Careggi BMT Unit Department of Haematology — http://www.aou-careggi.toscana.it/internet/index.php
- See also: Hospital Germans Trias i Pujol — http://www.gencat.net/ics/germanstrias/
- See also: Hospital Clinic of Barcelona — http://www.hospitalclinic.org/
- See also: Hospital de la Santa Creu i Sant Pau — http://www.santpau.es/
- See also: ULCA — http://www.ucla.edu/